CLINICAL TRIAL: NCT04214093
Title: A Phase I, Open-Label, Multicenter Study to Assess the Safety, Tolerability, Pharmacokinetics and Preliminary Antitumor Activity of Ascending Doses of AZD0466 in Patients With Advanced Hematologic or Solid Tumors
Brief Title: A Study of AZD0466 in Patients With Advanced Hematologic or Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Strategic change to clinical development plan
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D8240C00003; REFMAL 661 (Other: Sarah Cannon Development Innovations, LLC)
Record Dates: First submitted 2019-12-12; First posted 2019-12-30 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Advanced Solid Tumors; Lymphoma; Multiple Myeloma; Hematologic Malignancies
Keywords: AZD0466; Advanced solid tumors; Relapsed, refractory hematologic malignancies; Multiple myeloma; Tumor lysis syndrome
MeSH Terms: conditions — Lymphoma; Multiple Myeloma; Hematologic Neoplasms; Recurrence; Tumor Lysis Syndrome | interventions — AZD0466

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Dose escalation for patients with solid tumors, lymphoma and multiple myeloma with low risk of TLS. Each cohort within Arm A will test a single dose level.
  Interventions: Drug: AZD0466
- Arm B (Experimental): Dose escalation for patients with hematologic malignancies with an intermediate to high risk of TLS. Intrapatient dose ramp-ups within each cohort will be used.
  Interventions: Drug: AZD0466

INTERVENTIONS:
Drug: AZD0466 — In Arm A, AZD0466 will initially be administered IV over one hour, once weekly to the first cohort of patients. Subsequent cohorts of patients within Arm A are planned to receive sequentially higher doses.
  In Arm B, intrapatient dose ramp-ups will involve beginning at a specified starting dose and weekly increasing the dose to a maximum target dose for the cohort.

SUMMARY:
This is a first-time-in-human (FTIH), Phase 1 study to determine the safety, tolerability, maximum tolerated dose (MTD), recommended Phase 2 dose (RP2D), and pharmacokinetics (PK) of AZD0466 in patients with solid tumors, lymphoma and multiple myeloma at low risk for tumor lysis syndrome (TLS), as well as in patients at intermediate risk or high risk of TLS with hematologic malignancies for whom no standard therapy exists. Once an MTD/RP2D has been determined in the dose escalation portion, further disease-specific expansions (solid tumor and hematologic) will be undertaken. Combinations of AZD0466 with other standard of care treatments may be evaluated in the future.

DETAILED DESCRIPTION:
This is a FTIH study designed to evaluate the safety and tolerability of AZD0466 at increasing doses in patients with malignancies for whom no standard therapy exists, including advanced solid tumors, lymphoma and multiple myeloma with a low risk for TLS (Arm A), and relapsed, refractory hematological malignancies with an intermediate to high risk of TLS (Arm B). The study will also characterize the PK of AZD0466 and explore potential biological activity by assessing pharmacodynamics, exploratory biomarkers, and anti-tumor activity. Once an MTD/RP2D has been determined during escalation, further disease-specific expansions, possibly including, but not limited to small cell lung cancer, acute lymphoblastic leukemia, and acute myeloid leukemia will begin.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated written informed consent prior to any study specific procedures, sampling and analyses
2. Documented active disease requiring treatment that is relapsed or refractory as determined by RECIST or clinically defined changes.
3. Aged ≥18 yrs
4. Eastern Cooperative Oncology Group (ECOG) performance status ≤1 without 2 levels of ECOG deterioration within 2 weeks (wks) of signing the ICF
5. Life expectancy ≥12 wks
6. Measurable or evaluable disease according to disease-specific tumor assessment criteria
7. Adequate hepatic/renal function at screening:

   * AST and ALT ≤2.5 x Upper Limit of Normal (ULN)
   * Bilirubin ≤1.5 x ULN (unless bilirubin rise is due to Gilbert's syndrome or is of non-hepatic origin)
   * Creatinine ≤1.5 x ULN and creatinine clearance (CrCl) ≥50 mL/min, measured or calculated by Cockgroft-Gault method
8. Adequate cardiac function demonstrated by left ventricular ejection fraction ˃50% on screening echocardiogram
9. International normalized ratio ˂1.2 x ULN
10. Lipase ≤1.5 x ULN and serum amylase ≤1.5 x ULN and no prior history of pancreatitis
11. Patient agrees to the collection of formalin fixed paraffin embedded block or slides from archival diagnostic samples or a pre-treatment tumor biopsy
12. Willing and able to participate in all required study evaluations and procedures including receiving IV administration of study drug and admission to the hospital, when required, for at least 24 hrs during administration of study drug
13. Women should use adequate contraceptive measures, should not breast feed and should have a negative pregnancy test prior to start of dosing, or must have evidence of non-child-bearing potential by one of the following criteria at screening:

    * Women ˂ 50 yrs would be considered postmenopausal if they have been amenorrhoeic for the last 12 months following the cessation of exogenous hormonal treatments, and have serum follicle-stimulating hormone and luteinizing hormone levels in the postmenopausal range for the institution
    * Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation
14. Men should be willing to use barrier contraception (i.e., condoms) and refrain from sperm donation during and after the conduct of the trial

Inclusion Criteria for Arm A low risk of TLS (dose escalation):

1. Patient has histologically or cytologically confirmed diagnosis or an advanced, unresectable and/or metastatic malignancy for which there are no treatment options available known to provide clinical benefit as follows: Solid tumor, Lymphoma that meets TLS low risk criteria, Multiple myeloma
2. Adequate hematologic function independent of transfusion and growth factor support for ≥7 days before screening assessment. Solid tumors/lymphoma/multiple myeloma without bone marrow (BM) involvement:

   * Absolute neutrophil count ≥1,000 cells/mm^3
   * Hemoglobin ≥9.0 g/dL
   * Platelet count ≥100,000 cells/mm^3, or ≥35,000 cells/mm^3 with BM involvement

Inclusion Criteria for Arm B intermediate risk (IR) and high risk (HR) TLS (dose escalation):

1. Patients with histologically confirmed, relapsed or refractory hematologic malignancy for which there are no treatment options available known to provide clinical benefit. Patients must be classified as IR or HR TLS.
2. Adequate hematologic function independent of transfusion and growth factor support for ≥7 days before screening assessment
3. For AML and CMML patients, WBC must be ˂15,000/µL. Treatment with hydroxyurea (HU) prior to study entry and during ramp-up to achieve this level is permitted, as long as there is ˃24 hrs between the start of study drug and use of HU.
4. ALL/AML/MDS (IPSS-R intermediate/high/very high) and patients with BM involvement:

   * No hematologic inclusion criteria
   * Patient should be responsive to platelet transfusions to a minimum of 25,000 cells/mm^3 and having no history of thrombocytopenic bleeding

Exclusion Criteria

1. Patient has non-secretory myeloma
2. Patient has idiopathic thrombocytopenic purpura
3. Previously refractory to platelet transfusion within 1 yr
4. Treatment with any of the following:

   * Most recent radiotherapy ˂ 3 wks prior to first study treatment
   * Treated with hormonal therapy, immunotherapy, chemotherapy or investigational drugs within ≤21 days or 5 half-lives (whichever is shorter) from enrollment
   * Major surgery (excluding placement of vascular access) ≤21 days from beginning of the study drug or minor surgical procedures ≤7 days.
   * Treatment with hematopoietic colony stimulating factors (e.g., filgrastim, sargramostim) within 7 days of the first dose of study drug, or pegfilgrastim or darbepoetin within 14 days of the first dose of study drug
   * Patient has prescription/non-prescription drugs or other products known to be sensitive BCRP, OCT2, OAT3, OAT P1B1, OAT P1B3, CYP2B6, CYP2C8, CYP2C9, or CYP 2D6 substrates, or reversible strong and moderate CYP3A inhibitors, which cannot be discontinued within 5 half-lives of the drug before Day 1 of dosing and withheld throughout the study until 14 days after the last dose of AZD0466
   * Co-administration of CYP3A4 strong and moderate mechanism-based inhibitors or inducers which cannot be discontinued within 5 half-lives plus 12 days of the drug before Day 1 of dosing and withheld until 14 days after the last dose of AZD0466
   * Concurrent anti-coagulation therapy including aspirin which cannot be stopped
   * History of medications with known risk of Torsades de Pointes (cardiac arrhythmia due to drug-induced QTc prolongation) ≤5 half-lives before the start of treatment and continuing until 5 half-lives after the last dose of AZD0466
   * The use of live attenuated vaccines during the study through 30 days after the last dose of study drug
5. All toxicities from prior cancer therapy greater than NCI-CTCAE Grade (Gr) 1 will have returned to Gr1 at the time of enrollment with the exception of alopecia. Patients with Gr≤2 neuropathy are eligible.
6. Previously untreated brain metastases. Patients who have received radiation or surgery for brain metastases are eligible if therapy was completed at least 21 days previously and there is no evidence of CNS disease progression or mild neurologic symptoms.
7. Presence or history of CNS lymphoma, leptomeningeal disease or spinal cord compression
8. Active infection including HIV, Hepatitis B, or Hepatitis C
9. As judged by the Investigator, any evidence of severe or uncontrolled systemic diseases, (e.g., severe hepatic impairment, interstitial lung disease [bilateral, diffuse, parenchymal lung disease]); current unstable or uncompensated respiratory or cardiac conditions; uncontrolled hypertension; history of, or active, bleeding diatheses (e.g., hemophilia or von Willebrand disease); uncontrolled active systemic fungal, bacterial, viral, or other infection (exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics/other treatment); or IV anti-infection treatment within 14 days before first dose of study drug
10. Patients who have a high risk of developing renal dysfunction/renal involvement
11. Undergone any of the following procedures or experienced any of the following conditions currently or in the preceding 6 months:

    * Coronary artery bypass graft
    * Angioplasty
    * Vascular stent
    * Myocardial infarction
    * Angina pectoris
    * Congestive heart failure (New York Heart Association Class ≥2)
    * Ventricular arrhythmias requiring continuous therapy
    * Supraventricular arrhythmias, including atrial fibrillation, which are uncontrolled
    * Hemorrhagic or thrombotic stroke, including transient ischemic attacks or any other CNS bleeding
12. Any of the following cardiac criteria:

    * History of cardiomyopathy, myocarditis, or heart failure
    * Mean resting corrected QT interval (QTcF) ≥470 msec obtained from 3 ECGs in the absence of a cardiac pacemaker
    * Any clinically important abnormalities in rhythm, conduction, or morphology of resting ECG (e.g., complete left bundle branch block, third degree heart block, intermittent or persistent bundle branch block, AV block II-II or clinically significant sinus pause)
    * Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalaemia, congenital long QT syndrome, or family history of long QT syndrome or unexplained sudden death under 40 yrs of age
13. Abnormal ECHO at screening LVEF ≤50%
14. History of hypersensitivity to polyethylene glycol (PEG), PEGylated products or drugs with a similar chemical structure or class to AZD0466 or other BH3 mimetic
15. Lactating, breastfeeding, or positive pregnancy test
16. Patient has a prior history of another life-threatening malignancy ≤2 yrs prior to first dose of study drug with the exception of:

    * Malignancy treated with curative intent and with no evidence of active disease present for more than 2 yrs before screening and felt to be at low risk of recurrence by the treating physician
    * Adequately treated lentigo malignant melanoma without current evidence of disease or adequately controlled non-melanomatous skin cancer
    * Adequately treated carcinoma in situ without current evidence of disease
17. Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol
18. Judgement by the Investigator or Medical Monitor that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions, and requirements

Exclusion criteria for Arm A low risk of TLS (dose escalation):

1. Patients at IR or HR of developing TLS, including:

   * T-cell, diffuse large B-cell, peripheral T-cell, transformed, and mantle cell (blastoid variants) lymphoma patients with LDH ˃ULN
   * Early and advanced stage Burkitt lymphoma or lymphoblastic lymphoma patients
   * ALL, CLL, Richter's syndrome, AML, AML secondary, MDS, and chronic myelomonocytic leukemia (CMML)
2. Patients with a low risk of TLS that have significant renal dysfunction and/or renal involvement. Patients with CrCl ˂80 mL/min and/or who have higher tumor burden may be handled as TLS IR or HR patients.

Exclusion criteria for Arm B IR and HR TLS (dose escalation):

1. Patients with hematologic malignancies at HR of developing TLS are excluded from the first three cohorts. This includes:

   * ALL patients with white blood cell (WBC) counts ≥15 x 10^9/L with no HU in last 24 hrs or with WBC counts ˂100 x 10^9/L accompanied by LDH ≥2 x ULN
   * AML patients with WBC counts ≥100 x 10^9/L with no HU in the last 48 hrs
   * Patients with acute Burkitt leukemia
2. Patients with IR disease for TLS that also exhibits significant renal dysfunction, i.e., CrCl as calculated by Cockcroft-Gault method, if classified at investigator discretion as high-risk

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-12-16 (Actual); Primary Completion 2021-06-18 (Actual); Study Completion 2021-06-18 (Actual)

PRIMARY OUTCOMES:
The incidence of Dose Limiting Toxicities (DLTs) | 28 days for Arm A; between 35 and 56 days for Arm B due to varying number of ramp-up doses
  The maximum tolerated dose (MTD) will be determined by assessing the incidence of DLTs.
The incidence of adverse events | Minimum observation period 28 days for Arm A and between 35 and 56 days for Arm B due to varying number of ramp-up doses; and will continue until the subject is off the study (approximately 6 months)
  Safety and tolerability will be assessed in terms of adverse events as measured by Common Terminology Criteria for Adverse Events (CTCAE) version 5.

SECONDARY OUTCOMES:
Characterize the pharmacokinetic profile of AZD4320 by estimating maximum plasma concentration (Cmax) | Plasma PK will be measured at each cycle throughout study treatment for approximately 6 months. Cylce length is 28 days for Arm A and between 28-56 days for Arm B due to varying number of ramp-up doses.
  AZD0466 exposure is evaluated indirectly by AZD4320 concentration measurement. Total AZD4320 is the sum of dendrimer conjugated AZD4320 and released AZD4320. Released AZD4320 in the plasma is the sum of protein bound and unbound AZD4320 which is not dendrimer conjugated.
Characterize the pharmacokinetic profile AZD4320 by estimating area under the plasma concentration-time curve (AUC) | Plasma PK will be measured at each cycle throughout study treatment for approximately 6 months. Cycle length is 28 days for Arm A and between 28-56 days for Arm B due to varying number of ramp-up doses.
  AZD0466 exposure is evaluated indirectly by AZD4320 concentration measurement. Total AZD4320 is the sum of dendrimer conjugated AZD4320 and released AZD4320. Released AZD4320 in the plasma is the sum of protein bound and unbound AZD4320 which is not dendrimer conjugated.
Characterize urine pharmacokinetic profile of AZD4320 by renal clearance | Urine PK will be measured up to 48 hrs after the first treatment dose for select cohorts in Arm A, and pre-infusion and up to 48 hrs after the target dose for select cohorts in Arm B.
  AZD0466 exposure is evaluated indirectly by AZD4320 concentration measurement. Total AZD4320 is the sum of dendrimer conjugated AZD4320 and released AZD4320. Released AZD4320 in the plasma is the sum of protein bound and unbound AZD4320 which is not dendrimer conjugated.
Characterize urine pharmacokinetic profile of AZD4320 by amount excreted unchanged | Urine PK will be measured up to 48 hrs after the first treatment dose for select cohorts in Arm A, and pre-infusion and up to 48 hrs after the target dose for select cohorts in Arm B.
  AZD0466 exposure is evaluated indirectly by AZD4320 concentration measurement. Total AZD4320 is the sum of dendrimer conjugated AZD4320 and released AZD4320. Released AZD4320 in the plasma is the sum of protein bound and unbound AZD4320 which is not dendrimer conjugated.
Number of patients with a tumor response | Every 2 cycles (approximately 8 wks) from initiation of study treatment for up to approximately 6 months.
  Disease-specific criteria will be used to assess tumor response.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Research Site, New Haven, Connecticut
  - Research Site, Boston, Massachusetts
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Nashville, Tennessee
  - Research Site, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Results of this clinical trial are available on www.astrazenecaclinicaltrials.com — https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Search
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8240C00003&attachmentIdentifier=212396ef-db8a-4e0c-9c1a-e0a7d18ee9b5&fileName=D8240C00003_redacted_CSR_Synopsis.pdf&versionIdentifier=